CLINICAL TRIAL: NCT06884150
Title: fNIRS-based Analysis and Evaluation of the Effect of Schroth Rehabilitation on Motor Functions in Adolescent Idiopathic Scoliosis (AIS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Kadriye Tombak, PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Akdeniz UniversityTombak
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
Keywords: fNIRS
MeSH Terms: conditions — Scoliosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Group 1: Control Group (healthy participants) Group 2: Scoliosis group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 15 participant, healthy
- Scoliosis group (Experimental): * Being between the ages of 8-16,
  * Being diagnosed with adolescent idiopathic scoliosis,
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participating in schroth exercises for 45 minutes, 2 days a week after receiving the relevant diagnosis
  Arms: Scoliosis group

SUMMARY:
This study investigates the effects of Schroth-based rehabilitation on cortical dynamics, body awareness, and quality of life in individuals with Adolescent Idiopathic Scoliosis (AIS). Using fNIRS technology, motor control processes will be monitored, and the impact of rehabilitation on brain activity will be assessed.

A total of 30 participants (15 healthy and 15 with AIS), aged 8-16, will be examined, with pre- and post-rehabilitation comparisons. Measurements will include static posture, Y-Balance Test, Schroth walking, and brain activity recordings. SPM analysis will be used to assess brain signals, and quality of life and cosmetic deformity perception will be statistically evaluated.

The findings will contribute to the integration of neuroimaging into rehabilitation assessment, helping to develop more effective treatment strategies.

DETAILED DESCRIPTION:
The evaluation of body schema and perception in the cortex of adolescent idiopathic scoliosis and the analysis of changes in brain regions functionally related to motor control and coordination between controls and the analysis of their developmental process with rehabilitation are very important in terms of contributing to the planning of a better effective rehabilitation process, increasing the patient's quality of life and evaluating the status of body representation related to the disease, its development and sustainability in daily life.

fNIRS-based postural control neuroimaging and analysis will provide pioneering information about body schema, postural balance, motor activation and their rehabilitation-oriented changes and brain plasticity, which will provide separate analysis of dynamic and static balance.

The changes created by body schema and perception in the cortex in individuals with AIS and the rehabilitation-oriented developmental process will be evaluated with functional near-infrared spectroscopy (fNIRS) solutions, specifically in motor control and coordination.

Another important deficiency in the literature is the evaluation of changes created by rehabilitation processes in the cortex. Thanks to neural plasticity, a system that tries to compensate for a dysfunction can be reorganized. Therefore, rehabilitation studies are also of great importance here. The observed significant lateralization and body schema changes may also be useful for creating personalized and targeted corrective postural exercises.

The portable fNIRS device is an effective neuroimaging and analysis method for monitoring motor control processes in cortical areas in subjects moving without any movement restrictions. Therefore, especially in terms of body representation, since performing measurements in a limited area where the patient's movement is not possible, such as fMRI, does not provide very accurate results, especially since the evaluation of the change process created by motor movements in the cortex does not yield very accurate results, cortical dynamics in AIS individuals will be evaluated with fNIRS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 8-20
* Being diagnosed with adolescent idiopathic scoliosis,
* Accepting voluntary participation in the study.

Exclusion Criteria:

* History of tumor, vertebral malformation, trauma, epilepsy,
* Having had spine or lower extremity surgery,
* Having diagnosed psychiatric problems,
* Having any disease that would prevent them from exercising,
* Having rheumatic disease,
* Having congenital deformity,
* Being on another treatment for scoliosis during the study period,
* Having received any conservative treatment for scoliosis or posture disorder in the last six months,
* Having a body mass index over 25,

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
fNIRs device | Between 3th month-9th month
  After the installation and testing of the FNIRS device, recording and analysis are performed.
Y-balance test | Between 3th month-9th month
  Determination of maximum percentage reach and combined score from the Y-balance test,

SECONDARY OUTCOMES:
Scoliosis Research Society-22 (SRS-22) | Between 3th month-9th month
  Quality of life scale is determined with 5 sub-scores and a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
A consent form will be obtained from the individuals participating in the study or their parents.
Supporting Information: ICF
Time Frame: Between 3th month-9th month

REFERENCES:
- [Background] Surgent OJ, Dadalko OI, Pickett KA, Travers BG. Balance and the brain: A review of structural brain correlates of postural balance and balance training in humans. Gait Posture. 2019 Jun;71:245-252. doi: 10.1016/j.gaitpost.2019.05.011. Epub 2019 May 6. PMID 31082657
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31082657/